CLINICAL TRIAL: NCT04054440
Title: Outpatient Office Based Endovascular Procedures
Status: Enrolling by invitation | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 020.VSX.2013.D
Record Dates: First submitted 2019-08-12; First posted 2019-08-13 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Chronic Venous Insufficiency; Peripheral Arterial Disease; Dialysis Access Malfunction; Arterio-venous Fistula; Thoracic Outlet Syndrome; Vertebral Artery Insufficiency; Varicose Veins
Keywords: office based angiosuite
MeSH Terms: conditions — Peripheral Arterial Disease; Arteriovenous Fistula; Thoracic Outlet Syndrome; Vertebrobasilar Insufficiency; Varicose Veins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The results of this study will serve as a starting point for future trials concentrating on the effectiveness and clinical outcomes of the procedures performed in an office based angiosuite. Additionally, other studies could compare clinical outcomes between procedures performed in an office based angiosuite and other settings.

DETAILED DESCRIPTION:
Endovascular surgery combined with the demands of patients and physicians for less invasive procedures, have make this type of surgery one of the most innovative fields in medicine. However the endovascular experience in an office-based angiosuite is different from that in a hospital suite, and has been viewed in the past by some physicians as unsafe because it lacks the safety net of immediate hospital resources. In 2005, medicine allowed endovascular procedures to be performed in the office setting. The results of this study will serve as a starting point for future trials concentrating on the effectiveness and clinical outcomes of the procedures performed in an office based angiosuite.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Diagnosis of peripheral arterial disease (PAD), chronic venous insufficiency, dialysis access and malfunctioning arteriovenous fistulas, varicose veins, vertebrobasilar insufficiency, and thoracic outlet syndrome.
* Procedures performed as an outpatient in an office based angiosuite.

Exclusion Criteria:

* Age ≤ 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients who received endovascular procedures performed by board certified vascular surgeons in office-based angiosuites, located in California and Texas.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-06-20 (Actual); Primary Completion 2024-05-17 (Estimated); Study Completion 2024-05-17 (Estimated)

PRIMARY OUTCOMES:
Discharge location | April 2006 to December 2018
  classified as home, hospital floor, ICU and emergency room.
postoperative complications | April 2006 to December 2018
  events that disrupted the normal recovery process of the patient within the 24 hours following the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Sam S Ahn, MD, Principal Investigator — DFW Vascuclar
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States